CLINICAL TRIAL: NCT01622400
Title: Randomized Prospective Trial Evaluating the Efficacy of a Dedicated Therapeutic Education Program on the Blood Pressure and Other Cardiovascular Risk Factors Control in General Practice Patients at High Cardiovascular Risk
Brief Title: Efficacy of a Dedicated Therapeutic Education Program in Patients at High Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Association HTA Vasc (Other); CRESGE (Centre de Recherches Economiques Sociologiques et de Gestion) (Unknown); CERIM (Centre d'Etudes et de Recherche en Informatique Médicale), P. Devos (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-34; 2011-A00333-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2011-10-24; First posted 2012-06-19 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: High Blood Pressure
Keywords: Cardiovascular risk, Therapeutic education, General practice
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic education HTA Vasc (Experimental): 125 subjects who participate in the therapeutic education program
  Interventions: Other: Therapeutic education HTA Vasc
- Control group (No Intervention): 125 subjects who don't participate in the therapeutic education program

INTERVENTIONS:
Other: Therapeutic education HTA Vasc — The intervention program takes place in 3 phases. First, the education team realizes an individual educational diagnosis to define the objectives of the intervention according to each patient's needs. Secondly, patients assist to 3 to 5 group sessions lasting 2 hours with a dedicated nurse focusing on medical therapy explanation and blood pressure self measurement education - and with a dedicated nutritionist focusing on stress management and nutrition program. Patients can also have individual consultations with the dedicated nutritionist. Finally, an individual assessment permits to evaluate the benefits of the program for each patient and to define new objectives.
  Other Names: Program proposed by the association HTA Vasc
  Arms: Therapeutic education HTA Vasc

SUMMARY:
A dedicated therapeutic education program is an essential tool in the management of hypertension as well as in the control of other cardiovascular risk factors. The purpose of this study is therefore to evaluate the effect of such a therapeutic education program in general practice patients at high cardiovascular risk.

DETAILED DESCRIPTION:
Current guidelines for the prevention of cardiovascular disease recognize the major interest of an optimal control of all cardiovascular risk factors. It includes high blood pressure reduction, dietetic measures (weight loss - control of dyslipidemia and diabetes - regular physical activity), smoking cessation, stress management, … In that way, some authors suggest that it is essential for patients at high risk to have knowledge about their own pathology, medication, and to better understand the real benefit of specific lifestyle behaviors and the importance of blood pressure and glycaemia surveillance … The aim of this randomized controlled trial is to evaluate the efficacy of a dedicated therapeutic education program to control blood pressure and other cardiovascular risk factors in general practice patients at high cardiovascular risk.

250 patients are being enrolled. All patients will receive standard care but only 125 patients (randomized 1 to 1) will receive a structured therapeutic education program.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman of more than 18 years with a health insurance policy
* General practice patients who are agree to participate of the program of patient's therapeutic education in Lille (59) or Arras (62)
* Written informed consent must be obtained prior to performing any study-specific procedures
* Patient at high cardiovascular risk (Patient with a high blood pressure and 3 cardiovascular risk factors and/or Patient with cardiovascular disease)

Exclusion Criteria:

* Patient unwilling to take part to the therapeutic education program or to the study
* Patient not suitable to participate in the therapeutic education program
* Patient with dementia
* Anticipated survival (due to comorbidities) of less than one year from baseline
* Patient with current addiction or current alcohol / drug abuse
* Patient with known plans to move to another area of the country
* Unable to obtain written informed consent
* Patient who are pregnant or lactating
* Person without liberty by administrative or judiciary decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
High Blood Pressure in 12 months | 12 months
  Percentage of patients with a blood pressure of 140/90 mmHg or less in 12 months

SECONDARY OUTCOMES:
High Blood pressure at 24 months | 24 months
  Percentage of patients with a blood pressure of 140/90 mmHg or less in 24 months

CONTACTS AND LOCATIONS:
Overall Officials: FAYOLLE PF Patrick, GP, Principal Investigator — Arras Principal Investigator; GOUDJI GG Gustave, GP, Principal Investigator — Lille Principal Investigator
Locations (2):
- France (2):
  - General Practice Office, Arras
  - General practice office, Lille